CLINICAL TRIAL: NCT04582669
Title: Optimizing Intralesional Triamcinolone Dosing for Hidradenitis Suppurativa
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was administratively closed.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-12227
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Sodium Chloride 0.9% (Placebo Comparator): Each active hidradenitis suppurativa lesion will be injected with up to 1 mL of sodium chloride 0.9% in up to 3 anatomic areas. The maximum treatment volume is 3 mL.
  Interventions: Drug: Placebo
- Intralesional Triamcinolone 10 mg/mL (Active Comparator): Each active hidradenitis suppurativa lesion will be injected with up to 1 mL of intralesional triamcinolone 10 mg/mL in up to 3 anatomic areas. The maximum treatment volume is 3 mL.
  Interventions: Drug: Intralesional Triamcinolone 10 mg/mL
- Intralesional Triamcinolone 20 mg/mL (Experimental): Each active hidradenitis suppurativa lesion will be injected with up to 1 mL of intralesional triamcinolone 20 mg/mL in up to 3 anatomic areas. The maximum treatment volume is 3 mL.
  Interventions: Drug: Intralesional Triamcinolone 20 mg/mL
- Intralesional Triamcinolone 40 mg/mL (Experimental): Each active hidradenitis suppurativa lesion will be injected with up to 1 mL of intralesional triamcinolone 40 mg/mL in up to 3 anatomic areas. The maximum treatment volume is 3 mL.
  Interventions: Drug: Intralesional Triamcinolone 40 mg/mL

INTERVENTIONS:
Drug: Intralesional Triamcinolone 10 mg/mL — Injection of 1 mL intralesional triamcinolone 10 mg/mL in up to 3 anatomic areas.
  Arms: Intralesional Triamcinolone 10 mg/mL
Drug: Intralesional Triamcinolone 20 mg/mL — Injection of 1 mL intralesional triamcinolone 20 mg/mL in up to 3 anatomic areas.
  Arms: Intralesional Triamcinolone 20 mg/mL
Drug: Intralesional Triamcinolone 40 mg/mL — Injection of 1 mL intralesional triamcinolone 40 mg/mL in up to 3 anatomic areas.
  Arms: Intralesional Triamcinolone 40 mg/mL
Drug: Placebo — Injection of 1 mL sodium chloride 0.9% in up to 3 anatomic areas.
  Arms: Sodium Chloride 0.9%

SUMMARY:
Currently, there is limited evidence showing increased resolution of HS flares with higher doses of intralesional triamcinolone (ILTAC) as well as a difference in side effect profile between the doses. The goal of this study is to determine the efficacy of treating HS flares with ILTAC-10, ILTAC-20 and ILTAC-40 and to investigate the side effect profile for each dose.

DETAILED DESCRIPTION:
A double-blinded, randomized, placebo-controlled study examining the relative efficacy of ILTAC-10, ILTAC-20, and ILTAC-40 versus placebo for acute flares of HS in subjects with moderate to severe HS. The duration of the study will be approximately 4 weeks for each enrolled patient and will include an initial screening/randomization/treatment visit and a 4-week follow-up period. During the initial visit, subjects who meet the study's eligibility criteria will be randomized to receive either ILTAC-10, ILTAC-20, ILTAC-40, or placebo in a 1:1:1:1 ratio. Study subjects will then receive treatment or placebo. The follow-up period will be of 4 weeks and will consist of 3 phone calls and 1 live visit, including an end of study visit on week 4 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age > 13 years old.
* Subject must voluntarily sign and date an informed consent, approved by an independent ethics committee / institutional review board.
* Subject is willing to comply with the procedures in this protocol.
* The subject must be diagnosed with HS and receiving care at HSC
* Subjects with Hidradenitis Suppurativa Physician Global Assessment (HS-PGA) score between 2 and 5
* The subject must have an inflamed nodule or abscess at the time of enrollment.

Exclusion Criteria:

* The subject has an HS-PGA score of 0 or 1
* The subject has received ILTAC less than 8 days prior to the initial visit.
* The subject does not have capacity to consent to the study.
* The subject is has taken systemic steroids at least 4 weeks prior to the time of enrollment.
* The subject has a known allergy or history of adverse reaction to steroids.
* The subject is pregnant.
* Subjects who have received a biologic therapy two weeks before and during the study period.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Cohen, MD, MPH, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Steven Cohen, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Started | 3 | 3 | 2 | 3
Completed | 2 | 2 | 0 | 1
Not Completed | 1 | 1 | 2 | 2
Not completed — Subject missed appointment(s). | 1 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL | Total
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 11
Age, Customized [Count of Participants; unit: Participants]
  Age 20-29 years old | 3 | 2 | 0 | 2 | 7
  Age 30-39 years old | 0 | 0 | 0 | 1 | 1
  Age 40-49 years old | 0 | 1 | 1 | 0 | 2
  Age 50-59 years old | 0 | 0 | 0 | 0 | 0
  Age 60-69 years old | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 1 | 1 | 0 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 2 | 0 | 0 | 1 | 3
  Caucasian | 0 | 0 | 0 | 0 | 0
  American Indian/Alaskan Native | 0 | 0 | 0 | 0 | 0
  Pacific Islander | 0 | 0 | 0 | 0 | 0
  Hispanic | 0 | 3 | 2 | 0 | 5
  Asian | 0 | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Numeric Rating Scale (NRS)
Description: Numeric Rating Scale is a pain scale scored with whole integers from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable". Higher score indicates worse pain.
Time Frame: Baseline, Days 2, 6, 14, and 28
Population: NRS scoring data was not collected and aggregated and/or analyzed at any of the identified timepoints.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Hidradenitis Suppurativa-Physician Global Assessment (HS-PGA) Score
Description: HS-PGA is a six-staged physician global assessment tool (score ranges from 0 to 5) based on number of HS lesions including inflammatory and/or non-inflammatory nodules, abscesses, and draining fistulas. Higher HS-PGA score indicates more severe HS disease.
Time Frame: Baseline and Week 4
Population: HS-PGA scoring data was not collected and aggregated and/or analyzed at any of the identified timepoints.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: CRP (measured in mg/dL) is an inflammatory marker. A higher value is correlated with more severe disease.
Time Frame: Baseline and Week 4
Population: CRP data was not collected and aggregated and/or analyzed at any of the identified timepoints. Laboratory analyses were not conducted.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Hidradenitis Suppurativa (HS) Lesion Size
Description: HS lesion size will be measured using a metric ruler in centimeters. Measurement will be standardized according to greatest diameter as lesions will be measured from edge of one border to the edge of the opposite border.
Time Frame: Baseline and Week 4
Population: HS lesion size data was not collected and aggregated and/or analyzed at any of the identified timepoints.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) is a set of person-centered outcome measures that assesses physical, mental, and psychosocial health in adults and children. Clinical measures of health outcome includes physical function, mobility, pain, fatigue, emotional stress, ability to participate in social roles, sleep-related impairment, depressive symptoms/sadness, anxiety/fear, and anger. The scores are rated on a scale from 0 to 100 with "0" being "best functioning" and "100" being "worst functioning".
Time Frame: Baseline, Days 2, 6, 14, and 28
Population: PROMIS data was not collected/aggregated and therefore not analyzed at any of the identified timepoints.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Subjects Reporting Thinning and/or Atrophy of the Skin, Acneiform Lesion(s), Capillary Dilation(s), and Dyschromia When Compared to Baseline.
Description: Evaluate the morphologic changes in participant's skin from baseline, specifically assessing
  1. Acneiform lesion(s) are characterized by papules and pustules resembling acne vulgaris
  2. Capillary dilation(s) are bright red lines on skin surface and appear as linear or wavy or serpiginous; classified as telangiectasia(s) and/or spider angiomas.
  3. Dyschromia refers to alteration in skin pigmentation and can involve both hyperpigmented or hypopigmented macules.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 3 | 3 | 2 | 3
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Subjects Reporting Thinning and/or Atrophy of the Skin, Acneiform Lesion(s), Capillary Dilation(s), and Dyschromia When Compared to Baseline.
Description: as for outcome 6
Time Frame: Day 2
Population: There were two fewer subjects than baseline because subject(s) did not present for visit and/or meet eligibility criteria, and data was not collected and/or analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 3 | 2 | 1 | 3
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Subjects Reporting Thinning and/or Atrophy of the Skin, Acneiform Lesion(s), Capillary Dilation(s), and Dyschromia When Compared to Baseline.
Description: as for outcome 6
Time Frame: Day 6
Population: There was one fewer subject than baseline because subject did not meet eligibility criteria, and data was not collected and/or analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 3 | 2 | 2 | 3
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Subjects Reporting Thinning and/or Atrophy of the Skin, Acneiform Lesion(s), Capillary Dilation(s), and Dyschromia When Compared to Baseline.
Description: as for outcome 6
Time Frame: Day 14
Population: There were four fewer subjects than baseline because subject(s) did not present for visit and/or meet eligibility criteria, and data was not collected and/or analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 2 | 2 | 0 | 3
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Subjects Reporting Thinning and/or Atrophy of the Skin, Acneiform Lesion(s), Capillary Dilation(s), and Dyschromia When Compared to Baseline.
Description: as for outcome 6
Time Frame: Day 28
Population: There were six fewer subjects than baseline because subject(s) did not present for visit and/or meet eligibility criteria, and data was not collected and/or analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 2 | 2 | 0 | 1
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: ESR (measured in mm/h), is a pro-inflammatory marker. Higher ESR levels are correlated with greater hidradenitis suppurativa disease activity and worse clinical outcome.
Time Frame: Baseline and Week 4
Population: ESR data was not collected/aggregated and therefore not analyzed at any of the identified timepoints. Laboratory analyses were not conducted.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Baseline Patient Satisfaction Likert Scale
Description: Likert scale is a rating system that is designed to measure participant's overall attitude and perception regarding one's health and hidradenitis suppurativa. The scores range from 1 to 5 with "1" being "very unsatisfied" to "5" being "very satisfied". Higher scores indicate higher satisfaction.
Time Frame: Baseline
Population: Patient satisfaction data was not collected/aggregated and therefore not analyzed.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Patient Satisfaction Likert Scale
Description: as for outcome 12
Time Frame: Days 2, 6, 14, and 28
Population: Change from baseline data for patient satisfaction was not collected/aggregated and therefore not analyzed at any of the identified timepoints.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Interleukin-6 (IL-6)
Description: IL-6 (measured in pg/mL), is a pro-inflammatory cytokine. Higher IL-6 levels are correlated with greater hidradenitis suppurativa disease activity and worse clinical outcome.
Time Frame: Baseline and Week 4
Population: IL-6 data was not collected/aggregated and therefore not analyzed at any of the identified timepoints. Laboratory analyses were not conducted.
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sodium Chloride 0.9% | Intralesional Triamcinolone 10 mg/mL | Intralesional Triamcinolone 20 mg/mL | Intralesional Triamcinolone 40 mg/mL
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT04582669/Prot_SAP_000.pdf